CLINICAL TRIAL: NCT04716829
Title: Study of the Efficacy of the LUNA-EMG System on Motor Function in the Management of Neurological Disorders.
Brief Title: LUNA-EMG to Enhance Motor Functions in Neurological Disorders
Acronym: LUNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: CHU Liège - Belgium (Unknown)
Responsible Party: Principal Investigator, Aurore Thibaut, PhD, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-372
Record Dates: First submitted 2021-01-19; First posted 2021-01-20 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: stroke; EMG; rehabilitation; physiotherapy; occupational therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LUNA-EMG (Experimental): The experimental group will receive 30 minutes of training with the LUNA-EMG for 12 weeks.
  Interventions: Device: LUNA-EMG
- Control (No Intervention): The control group will receive its rehabilitation care.

INTERVENTIONS:
Device: LUNA-EMG — The LUNA-EMG (Samcom) system is a robot that allows the evaluation of muscular strength through the recording of muscle activity (electromyography - EMG) in order to provide precise objective data on the patient's muscle function. In addition to the diagnostic aspect (evaluation of muscle strength, range of motion and proprioception), the LUNA-EMG robot allows the adaptation of movements during rehabilitation sessions according to the individually generated strength.
  Arms: LUNA-EMG

SUMMARY:
The aim of the present study is to evaluate the effects of training performed with the LUNA-EMG system to enhance motor functions of the upper limb in stroke This is a randomized open-label trial. Patients will be randomized into the intervention group (LUNA-EMG) or in the control group (standard care).

The effect of the training will be measured with the EMG, the upper limb motor function and the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Having signed the informed consent

Exclusion Criteria:

* Acute pain syndrome
* Severe cognitive deficits
* Risk of fracture or unconsolidated fracture
* Rigid joints (spasticity, severe osteoarthritis and arthritis) or unstable joints
* Severe ataxia and apraxia
* Epilepsy
* Pacemakers and similar implants
* Insufficient skin conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
muscular strength in mV | 12 weeks
  muscular strength will be measured with the EMG

SECONDARY OUTCOMES:
Fugl-Meyer | 12 weeks
  The scale evaluates motor capacities of the upper limb following a stroke. Scores range from 0 to 66 (the higher the better).
Modified Ashworth Scale | 12 weeks
  This scale measures spasticity. The results are scored from 0 to 4 (the higher the more spastic).
Lovett | 12 weeks
  This scale measures muscular strength. The scale ranges from 0 to 5 (the higher the better).

CONTACTS AND LOCATIONS:
Locations (1):
- CNRF, Tinlot, Liege, Belgium

IPD SHARING:
Plan to Share IPD: Undecided